CLINICAL TRIAL: NCT02312193
Title: Evaluation of the Signaling Path of Emiline1-TGFβ in the Myogenic Tone of Resistance Arteries in a Population of Normotensive and Hypertensive Subjects
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, MD, Ph, Neuromed IRCCS
Other Study IDs: LMB02
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Hypertension
Keywords: hypertension; myogenic tone
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Case: Hypertensive subjects
- Control: Normotensive subjects

SUMMARY:
Aim of this study is to enhance the knowledge of myogenic tone alterations in hypertensive patients and to better understand the mechanisms controlling the myogenic tone. Evaluations will be performed through ex vivo studies of peripheral arterioles in human adipose tissue from lumbar muscle, isolated from biopsies. This will allow investigators to evaluate the myogenic function in response to progressive blood pressure increases, in order to correlate myogenic function to arterial hypertension and to the molecular mechanisms already identified in the preclinical models.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 30 and 70 years of age
* Hypertensive patients: Patients with a previous diagnosis of hypertension
* Normotensive patients: subjects without story of hypertension
* Written informed consent

Exclusion Criteria:

* Severe hypertension (eg, systolic >180 mm Hg, diastolic >110 mm Hg)
* Manifested or suspected secondary hypertension (coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, pheochromocytoma)
* History of cardiac complications (previous acute myocardial infarction (AMI), unstabile angina, percutaneous transluminal coronary angioplasty (PTCA), coronary artery bypass grafting (CABG), congestive heart failure (NYHA II-IV))
* Diabetes mellitus
* Renal pathologies (creatinine clearance < 30 ml/min)
* Severe hepatic dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients hospitalized in the Department of Neurosurgery of the IRCCS Mediterranean Neurological Institute Neuromed, according to specific inclusion criteria and undergoing surgery for disc disease. Subjects included in the study will be normotensive and hypertensive patients. Approximately 70 subjects of both genders (35 normotensive, 35 hypertensive) aged between 30 and 70 years old will be included in the study. All the enrolled patients must have an indication for neurosurgical intervention.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Myogenic tone measured by micromyographic technique to evaluate small-artery morphology. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy